CLINICAL TRIAL: NCT01651143
Title: Double-blind, Randomized, 8-week Placebo-controlled, and 16-week Open-label Extension Study Investigating the Safety, Pharmacokinetics and Pharmacodynamics of SAR100842 Given Orally to Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: Proof of Biological Activity of SAR100842 in Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT12339; 2012-001369-34 (EudraCT Number); U1111-1127-2854 (Other: UTN)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — SAR-100842

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR100842 (Experimental): Core part: SAR100842 300 mg, oral administration twice daily, for 8 weeks
  Extension part: SAR100842 300 mg, oral administration twice daily, for 16 additional weeks
  Interventions: Drug: SAR100842
- Placebo (Placebo Comparator): Core part: Placebo (for SAR100842), oral administration twice daily, for 8 weeks
  Extension part: SAR100842 300 mg, oral administration twice daily, for 16 additional weeks
  Interventions: Drug: SAR100842; Drug: Placebo (for SAR100842)

INTERVENTIONS:
Drug: SAR100842 — Pharmaceutical form: tablets
  Route of administration: oral
Drug: Placebo (for SAR100842) — Pharmaceutical form: tablets
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

- To evaluate safety and tolerability of 8-week oral administration of SAR100842 in patients with diffuse cutaneous systemic sclerosis.

Secondary Objectives:

* To evaluate the pharmacodynamic effect of SAR100842 in patients with systemic sclerosis as measured by disease related biomarkers and Lysophosphatidic acid (LPA) receptor signaling markers in blood and skin;
* To explore the effect of SAR100842 on skin thickness in patients with systemic sclerosis as measured by the modified Rodnan Skin Score (mRSS);
* To explore the effect of SAR100842 on quality of life as measured by the Scleroderma Modified Health Assessment Questionnaire (SHAQ);
* To document long term safety of SAR100842 during the extension part.

DETAILED DESCRIPTION:
Core part: randomized, double-blind, placebo-controlled study - 8-week treatment Extension part for participants completing the core part: Open label non-controlled study - 16-week treatment

Each patient's participation in the study will be approximately 13 or 33 weeks depending on their participation in the extension part: up to 2 weeks of screening, 8 weeks of treatment in the core part, 1 to 30 days wash-out between core part and extension part , 16 weeks of treatment in the extension part and 3 weeks of follow up.

ELIGIBILITY:
Inclusion criteria :

- Patients who meet the American College of Rheumatology (ACR) criteria for systemic sclerosis with diffuse cutaneous involvement and <36 months since the onset of the first systemic sclerosis manifestation other than Raynaud's phenomenon and have a Modified Rodnan Skin Score (mRSS) ≥ 15 and an area of definite involvement of the dorsal forearm that is considered amenable to repeated 4mm skin biopsies.

Exclusion criteria:

1. Patients with high dose or unstable low dose immunosuppressive drugs, cytotoxic, anti-fibrotic or glucocorticoids drugs at least 4 weeks prior to screening
2. Serum creatinine > 2.0 mg/dL
3. Gastrointestinal involvement preventing oral administration of study drug
4. Severe cardiac and/or pulmonary disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability during the 8 week treatment period (core part): Number of patients reporting adverse events | Up to 8 weeks

SECONDARY OUTCOMES:
Change from baseline to Week 8 in biomarkers obtained from blood and skin | Day 1 and Week 8 (core part)
Change from baseline to Week 8 in Modified Rodnan Skin Score (mRSS) | Day 1 and Week 8 (core part)
Change from baseline to Week 8 in Scleroderma Health Assessment Questionnaire (SHAQ) score | Day 1 and Week 8 (core part)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (7):
  - Investigational Site Number 840006, Scottsdale, Arizona
  - Investigational Site Number 840003, Washington D.C., District of Columbia
  - Investigational Site Number 840004, Baltimore, Maryland
  - Investigational Site Number 840001, Boston, Massachusetts
  - Investigational Site Number 840002, Ann Arbor, Michigan
  - Investigational Site Number 840007, New Brunswick, New Jersey
  - Investigational Site Number 840008, Pittsburgh, Pennsylvania
- France (2):
  - Investigational Site Number 250003, Lille
  - Investigational Site Number 250001, Paris
- Investigational Site Number 380001, Milan, Italy
- Investigational Site Number 756001, Zurich, Switzerland
- United Kingdom (2):
  - Investigational Site Number 826001, London
  - Investigational Site Number 826002, Salford

REFERENCES:
- [Derived] Allanore Y, Distler O, Jagerschmidt A, Illiano S, Ledein L, Boitier E, Agueusop I, Denton CP, Khanna D. Lysophosphatidic Acid Receptor 1 Antagonist SAR100842 for Patients With Diffuse Cutaneous Systemic Sclerosis: A Double-Blind, Randomized, Eight-Week Placebo-Controlled Study Followed by a Sixteen-Week Open-Label Extension Study. Arthritis Rheumatol. 2018 Oct;70(10):1634-1643. doi: 10.1002/art.40547. Epub 2017 Nov 6. PMID 29732731